CLINICAL TRIAL: NCT04927689
Title: Evaluation of an Environmental Counsellor's Home Stay in Children Treated for Asthma or Allergic Rhinitis Via a Standardized Medical Questionnaire Randomized Controlled Superiority Trial in Parallel Arms, Multicentric (EvalPCE)
Acronym: EvalPCE
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC21_0186
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Category 3 Study (Non-interventional Research)
Keywords: Asthma; Allergic rhinitis; Environmental consultant
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of asthmatic children and children with allergic rhinitis at day 0 and 6 months after a home visit by an environmental consultant via standardized medical questionnaires.

DETAILED DESCRIPTION:
Asthma and allergic rhinitis are chronic diseases whose control is multifactorial (drug treatment, therapeutic education of the family and the child, consideration of a possible allergen...). When this control is not optimal, it leads to significant school absenteeism, pediatric emergency room visits and hospitalizations. Environmental conditions at home play a role in asthma exacerbations and poor control of allergic rhinitis in children. Mites, animal allergens, passive smoking, molds, cockroaches, household products, etc., are the main causes. The visit of a home environment advisor, who intervenes on medical prescription, makes it possible to evaluate the source of allergens and pollutants in the home and then to propose changes to the home. This position was created in France in 2009 by the Ministry of the Environment and is funded by the Agence Régional de Santé (ARS - Regional Health Agency). The few studies carried out to assess the effectiveness of a home visit by an environmental advisor on exacerbations of these diseases are contradictory: some show an improvement in the quality of life of asthmatic children after a home visit (via the average reduction in the number of days with symptoms/year) as well as a reduction in asthma-related morbidity thanks to a reduction in exposure to indoor allergens. Others have shown that it does not reduce the number of emergency room visits for asthma exacerbations. Furthermore, it would appear that targeted allergen avoidance measures do not reduce drug treatment in asthmatics who are already on optimal pharmacological treatment.

To our knowledge, there are no studies in France that use standardized medical questionnaires to assess disease control and quality of life before and after the visit of a home environmental consultant. For example, in Angers and Nantes, evaluation questionnaires are carried out with patients at 6 months and 1 year after a home visit, but the answers are not standardized and sometimes very subjective.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 18 years of age
* With asthma or allergic rhinitis
* For whom a home visit by an environmental consultant is prescribed

Exclusion Criteria:

* Parental refusal to participate in the study
* Poor understanding of the French language not allowing to fill in the questionnaire
* Asthmatic child under 7 years old or child with allergic rhinitis under 6 years old (questionnaires not validated below these ages)
* Patient concerned by a current request for relocation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient under 18 years of age with asthma or allergic rhinitis for whom a home visit by an environmental consultant is prescribed
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Quality of life of asthmatic children and children with allergic rhinitis | 6 months
  Assessment of the quality of life of asthmatic children and children with allergic rhinitis at day 0 and 6 months after a home visit by an environmental consultant via standardized medical questionnaires.

SECONDARY OUTCOMES:
Disease control, health care utilization and change in drug therapy | 6 months
  Assessment of disease control, health care utilization and change in drug therapy of asthmatic children and children with allergic rhinitis at day 0 and 6 months after a home visit by an environmental consultant via standardized medical questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: CARBALLIDO, Study Director — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).